CLINICAL TRIAL: NCT02628717
Title: Interferon/Ribavirin-Free Sofosbuvir Based Treatment Regimens In Patients With Advanced Liver Disease - Results Of A Real-Life Austrian Ribavirin-/Interferon Free Cohort (AURIC)
Brief Title: Interferon/Ribavirin-Free Sofosbuvir Based Treatment (AURIC)
Acronym: AURIC
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Peter Ferenci, Prof., Medical University of Vienna
Other Study IDs: I3MHCV
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Chronic Hepatitis C; Cirrhosis
Keywords: Hepatitis C; sofosbuvir; ledipasvir; daclatasvir; simeprevir
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- SOF/SMV: SOF/SMV 400mg/150mg QD 12-24 weeks
- SOF/DCV: SOF/DCV 400mg/60mg QD 12-24 weeks
- SOF/LDV: SOF/LDV 400mg/90mg QD 12-24 weeks
- treatment duration: 12 - 24 weeks

SUMMARY:
Since the availability of interferon free direct acting antivirals (DAA) the centers authorized to prescribed these drugs in Austria submitted their data to a central data base (AURIC) using treatment regimes without interferon and ribavirin in patients with advanced liver disease (F3/4)

DETAILED DESCRIPTION:
From end of 2013 303 HCV-monoinfected patients with advanced liver disease (F3/4) were treated with interferon (IFN)-free and RBV-free SOF-based regimens. During this period only 7 patients received additional RBV. These patients were not included in this analysis. Only patients who completed 12 weeks of treatment-free follow up until July 2015 were included in this analysis. In Austria, prescription of DAAs is restricted to specialized treatment centers. Data are obtained by 6 participating centers and submitted to the central database forming for of the Austrian Ribavirin- and Interferon-free cohort (AURIC). Incoming data are reviewed by the staff of the hepatitis study group of the Dept. of Medicine III, Medical university of Vienna.The treatment regimens consisted of SOF/DCV, SOF/SMV, and SOF/LDV. The duration of treatment was based on a response guided approach at the discretion of the treating physician (12 or 24 weeks).

Sixty six patients who had started therapy before August 2014 received SMV or DCV as part of a named patient program, SOF was prescribed. For the remaining patients all drugs were prescribed and paid for by the Austrian social insurance.

This study will investigate various aspects of treatment response to regimens containing direct-acting antiviral agents for the treatment of chronic hepatitis C:

Sustained virologic response (SVR) defined as undetectable HCV-RNA after 12 weeks of treatment free follow up

Virological breakthrough/relapse defined as reappearance of HCV on treatment/during follow up

Impact of viral kinetics on prediction of treatment efficacy: Viral load measured repeatedly (at baseline, on days 2,7,14,21,28,and than every 4 weeks until end of treatment) allows to study the rapidity of viral clearance. This parameter was used to assess whether length of treatment can be modified. Plasma HCV RNA levels were quantified by One Signal Amplification (Versant HCV RNA 3.0),

Adverse Event Recording (using standard GCP criteria)

Longterm outcome after SVR based on examining patients with SVR in six monh intervals. Examination will include liver sonography, elastography, routine blood chemistry including alpha1-fetoprotein

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 or older) being treated with antiviral HCV treatment regimens

Exclusion Criteria:

* other disease with poor prognosis (ie. metastatic cancer, heart failure)
* participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with fibrosis grade F3 or F4, age >18 years, with indication for antiviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 558 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with sustained virologic response (SVR) | 12 weeks treatment free follow up
  SVR is defined by the undetectability of HCV-RNA after 12 weeks of treatment free follow up

SECONDARY OUTCOMES:
On treatment predictability of SVR | 12/24 weeks of treatment + 12 weeks of follow up
  Virus testing at baseline, day 2,7,14,21,28, than every 4 weeks until SVR. Rapidity of viral clearance may be a useful parameter to determine the duration of treatment
Number of patients with liver events (Mortality, Hepatic decompensation, Variceal Bleeding,Hepatocellular Carcinoma, Need for Liver Transplantation) on longterm clinical outcome | 3 years
  regular clinical visits including laboratory test, fibroscan and sonography will be performed every six months after achieving SVR

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | treatment (12 to 24 weeks) +12weeks treatment free follow up
  adverse events will be recorded and graded

CONTACTS AND LOCATIONS:
Overall Officials: Harald Hofer, MD,Prof, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria